CLINICAL TRIAL: NCT06469450
Title: KF2023#1-Trial: Influence of Statin Intake on Cellular Readouts
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mikko Niemi (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Mikko Niemi, Professor, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KF2023#1
Record Dates: First submitted 2024-05-06; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pharmacodynamics
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atorvastatin (Experimental): atorvastatin 40 mg daily for 28 days
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — one 40 mg atorvastatin tablet once daily for 28 days

SUMMARY:
A majority of high-risk patients does not achieve their cholesterol target levels and most of these patients do not receive more effective combination therapy, which goes beyond statin monotherapy. Large interindividual differences in treatment outcomes have been observed for patients receiving statins. Statins block cholesterol synthesis and increase cellular low-density lipoprotein (LDL) uptake. Importantly, LDL uptake is highly divergent in individuals.The aim of this trial is to investigate how atorvastatin influences leukocyte readouts of LDL uptake and lipid storage in humans. The trial is a single-arm, open-label, interventional trial. A total of 15 healthy volunteers will receive 40 mg atorvastatin once a day for 4 weeks. The participants will provide blood samples before starting the atorvastatin intervention, each week when taking atorvastatin, and one week after the end of the intervention for the measurement of leukocyte readouts of LDL uptake and lipid storage.

ELIGIBILITY:
Inclusion Criteria:

1. a signed written informed consent
2. age 18-40 years
3. healthy, and
4. Accepted results from laboratory tests (blood haemoglobin, basic blood count and blood platelets, alanine aminotransferase, alkaline phosphatase, glutamyl transferase, creatinine, plasma potassium and sodium). Negative pregnancy test result (serum human chorionic gonadotropin) for women.
5. Fully vaccinated against COVID-19.

Exclusion Criteria:

1. significant disease
2. smoking
3. SLCO1B1 poor function genotype
4. oral contraception or other continuous medication
5. pregnancy, planning of pregnancy or breastfeeding
6. participating in a clinical trial less than 3 months ago
7. donating blood less than 3 months ago
8. marked obesity
9. anticipated difficulties in drawing blood samples
10. weight less than 45 kg
11. BMI less than 18.5 kg/m2 or
12. inadequate Finnish language skills

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lipid trafficking score LT-Mo | Baseline and once a week for 5 weeks
  The primary outcome measurement is the "lipid trafficking score LT-Mo" is a combination of LDL uptake and lipid droplet quantifications in monocytes.
  The participants provide blood samples before starting the atorvastatin intervention, each week when taking atorvastatin (4 times in total), and one week after the end of the intervention.

SECONDARY OUTCOMES:
Leukocyte LDL uptake | Baseline and once a week for 5 weeks
  Systematic quantification of leukocyte uptake of low-density lipoprotein (LDL). Leukocytes are exposed to fluorescently labelled LDL particles and internalized LDL particles are quantified with microscopy and automated image analysis. The specific readouts are overall fluorescent LDL intensity and the number of endosomal organelles filled with fluorescent LDL particles for monocyte and lymphocyte subpopulations.
Leukocyte lipid storage | Baseline and once a week for 5 weeks
  A systematic semi-automated approach is used to quantify cellular lipid droplets, dedicated storage organelles for lipids. Individual lipid droplets, their size and area are quantified in each cell and either used as individual readouts or combined with LDL uptake readouts to derive lipid trafficking scores.
Atorvastatin plasma concentration | Once a week during the 4 week atorvastatin treatment
  The plasma concentrations of atorvastatin and its metabolites will be quantified with liquid chromatography tandem mass spectrometry (LC-MS/MS) from plasma samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No